CLINICAL TRIAL: NCT03240315
Title: Establishment of Individualized Prediction System for Acute Exacerbation of Chronic Obstructive Pulmonary Disease Based on Cloud Platform
Brief Title: Personalized Prediction Strategy for Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Guangzhou Science and Technology Innovation Commission,China (Unknown)
Responsible Party: Principal Investigator, Fengyan Wang, Principal Investigator, Guangzhou Institute of Respiratory Disease
Other Study IDs: 201604020012; 2017YFC1310600 (Other Grant/Funding Number: Ministry of Science and Technology of the People's Republic of China)
Record Dates: First submitted 2017-07-31; First posted 2017-08-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma,sputum

GROUPS / COHORTS (2):
- COPD subjects: Subjects with GOLD stage I-IV COPD
- Healthy control subjects: Ages 40 to 90, with no history of lung disease and no history of acute illness or medication use within the past month.

SUMMARY:
This is a 3-year longitudinal study designed to establish a personalized prediction and prevention system for acute exacerbations of chronic obstructive pulmonary disease (AECOPD). Data will be prospectively collected from patients with chronic obstructive pulmonary disease (COPD) and healthy control participants, including clinical characteristics, pathophysiological parameters, etiological factors, and immunological information. These data will be analyzed using data mining approaches combined with Internet-based technologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients was diagnosed as COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines older than 40 years old.

  * A signed and dated written informed consent is obtained prior to participation.
  * Able to comply with the requirements of the protocol and be available for study visits over 3 years.

Exclusion Criteria:

* A COPD subject will not be eligible for inclusion in this study if any of the following criteria apply:

  * Known respiratory disorders, or disorders identified at screening/visit 1 (including identification on the first CT scan), other than COPD (e.g.: lung cancer, sarcoidosis, tuberculosis, lung fibrosis, cystic fibrosis)
  * Known history of significant inflammatory disease, other than COPD (e.g. rheumatoid arthritis and Lupus)
  * Known to be severely alpha-1-antitrypsin deficient
  * Has experienced a moderate or severe exacerbation (requiring oral corticosteroid, antibiotics or hospitalisation) within the last 4 weeks
  * Having undergone lung surgery (e.g. lung reduction, lung transplant)
  * Have cancer or have had cancer in the 5 years prior to study entry
  * Having received a blood transfusion in the 4 weeks prior to study start
  * Inability to walk
  * Taking part in a blinded drug study
  * Having therapy with systemic corticosteroids at inclusion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD subjects in China
Sampling Method: Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Establishment of prediction platform for COPD exacerbation | 3 years
  The patients with chronic obstruction pulmonary disease will be followed up at intervals of 3 months for 3 years by the Modified British Medical Research Council (mMRC) score scale,spirometric analysis, sputum smear,questionnaire and so on. An exacerbation of COPD was diagnosed according to GOLD guidelines. Time to the first acute exacerbation and average number of acute exacerbations per year in COPD subjects will be record.Research of AECOPD Risk factors based on complex network analysis.Identification and validation of COPD exacerbations risk stratification and predictive markers based on data mining.

SECONDARY OUTCOMES:
Developing new protein chips for AECOPD | 3 years
  Systemic and airway autoantibody profiles and cytokine profiles will be measured using commercial multiplex bead-based assay to screen out a set of ideal AECOPD-related markers.
Detection of immune repertoire in COPD/AECOPD | 3 years
  Immune status of COPD patients will be investigated by using the immune repertoire technique and its relationship with the pathophysiology of AECOPD will be identified.
Pathogenic microorganism and drug resistance monitoring for COPD exacerbation | 3 years
  Dynamics of pathogenic microorganism and drug resistance in natural course of COPD will be investigated by using the metagenome technique and the culture technique.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD/Ph.D, Study Director — Guangzhou Institute of Respiratory Health,The First Affiliated Hospital of Guangzhou Medical University,China
Locations (1):
- Guangzhou Institute of Respiratory Health,The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Feng S, Yang Y, Liang Z, Song A, Chen J, Guo Z, Chen Z, Miao C, Yang H, He W, Zhou Z, Drummond MB, Chen R, Wang F. Association Between Airway Mucus Plugs and Risk of Moderate-to-Severe Exacerbations in Patients With COPD: Results From a Chinese Prospective Cohort Study. Chest. 2025 Sep;168(3):627-638. doi: 10.1016/j.chest.2025.03.026. Epub 2025 Apr 8. PMID 40210091
- [Derived] Cass SP, Yang Y, Xiao J, McGrath JJC, Fantauzzi MF, Thayaparan D, Wang F, Liang Z, Long F, Stevenson CS, Chen R, Stampfli MR. Current smoking status is associated with reduced sputum immunoglobulin M and G expression in COPD. Eur Respir J. 2021 Feb 4;57(2):1902338. doi: 10.1183/13993003.02338-2019. Print 2021 Feb. No abstract available. PMID 32883677